CLINICAL TRIAL: NCT02692092
Title: HealthEast Community Hip and Knee Replacement Registry
Acronym: HEJR
Status: Recruiting | Type: Observational
Sponsor: HealthEast Care System (Other)
Responsible Party: Sponsor
Other Study IDs: 03 12 007R
Record Dates: First submitted 2014-01-29; First posted 2016-02-25 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Bone Fracture
Keywords: Complications; Arthroplasty, Hip Replacement; Arthroplasty, Knee Replacement
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Arthroplasty Patients: Any patient who has received a total hip or total knee arthroplasty at a healtheast acute care hospital.

SUMMARY:
HealthEast Care System began the first community-based joint replacement registry (HJRR) in the U.S. in 1991, and now has more than 30,000 total joints registered. The purpose of the HJRR is to maintain and improve the care of individuals undergoing joint replacement surgery by providing timely information to their surgeons and the broader orthopaedic community.

As it moves into the third decade, the HJRR is proud of its role in the development of the national American Joint Replacement Registry (AJRR) and will remain an important contributor to the larger national effort in the advancement of orthopaedic science.

DETAILED DESCRIPTION:
HealthEast Care System began the first community-based joint replacement registry (HJRR) in the U.S. in 1991, with a database that allowed tracking of implant use and failure rates among the 90 orthopaedic surgeons performing arthroplasty surgery in the greater metropolitan area of St. Paul, MN. Initially conceived as part of a process to better manage costs and determine which implants were most cost-efficient, it became apparent that the registry would allow insight into the same process that had proven its value in the Scandinavian joint registries. With the knowledge that a majority of total joint arthroplasties in the U.S. are performed by relatively low-volume community surgeons, the HJRR remains uniquely positioned to reflect contemporary U.S. surgical practices.

The purpose of the HJRR is to maintain and improve the care of individuals undergoing joint replacement surgery by providing timely information to their surgeons and the broader orthopaedic community. With the primary outcome measure of time to revision surgery, combined with analysis of confounding factors and mortality monitoring, the HJRR can provide some realistic measure of the success of a given arthroplasty procedure in our community. In addition, the registry can evaluate the relative effectiveness of different prosthetic designs, identify patient variables that may impact implant survival, and provide the tracking mechanism necessary in the event of implant recalls.

Over the 20 years of its existence, the HJRR has refined its data-gathering, data verification, and data analysis and utilizes a process design that requires no direct surgeon involvement with data input. Volunteer surgeons review each revision chart and operative note to carefully delineate the reason for revision. The HJRR capture process has been validated and more than 94% of the revision surgery is performed within the HJRR. The database is used to generate information of practical use to the surgeon, and has been demonstrated to influence surgeon behavior. Among other examples, HJRR reports on the failure rates associated with unicompartmental knee arthroplasty, hybrid and cementless total knee arthroplasty, and metal-on-metal total hip designs have led to significant declines in their respective use over the periods documented. Similarly, the HJRR allowed for rapid notification of surgeons and expedited patient care during the three significant hip implant recalls of the last decade.

As it moves into the third decade, the HJRR is proud of its influential role in the development of the national American Joint Replacement Registry (AJRR) as one of the earliest participants and pilot hospitals. It will remain an important contributor to the larger national effort, particularly for certain data subsets that may be outside of the scope of the much larger AJRR. The HJRR core workgroup has published widely on its findings in the last two decades, and looks forward to the future as a compelling example of how worthwhile information and advancements in orthopaedic science can be made in the community setting.

ELIGIBILITY:
Inclusion Criteria:

* Total Hip or Total Knee Arthroplasty
* HealthEast acute care hospital

Exclusion Criteria:

* Age<18
* Primary procedure not performed at a HealthEast hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having total hip or knee arthroplasty at a HealthEast acute care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 1991-09; Primary Completion 2091-08 (Estimated); Study Completion 2091-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative Revision Rate | 10 Years
  Our end point of interest was revision for any reason, with revision defined as removal, exchange, or addition of components, requiring a second surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Terence J Gioe, MD, Principal Investigator — HealthEast Care System
Locations (1):
- HealthEast Care System, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gioe TJ, Sinner P, Mehle S, Ma W, Killeen KK. Excellent survival of all-polyethylene tibial components in a community joint registry. Clin Orthop Relat Res. 2007 Nov;464:88-92. doi: 10.1097/BLO.0b013e31812f7879. PMID 17589363
- [Result] Gioe TJ, Killeen KK, Mehle S, Grimm K. Implementation and application of a community total joint registry: a twelve-year history. J Bone Joint Surg Am. 2006 Jun;88(6):1399-404. doi: 10.2106/JBJS.E.01198. No abstract available. PMID 16757777
- [Result] Gioe TJ, Killeen KK, Grimm K, Mehle S, Scheltema K. Why are total knee replacements revised?: analysis of early revision in a community knee implant registry. Clin Orthop Relat Res. 2004 Nov;(428):100-6. PMID 15534527
- [Result] Gioe TJ, Killeen KK, Hoeffel DP, Bert JM, Comfort TK, Scheltema K, Mehle S, Grimm K. Analysis of unicompartmental knee arthroplasty in a community-based implant registry. Clin Orthop Relat Res. 2003 Nov;(416):111-9. doi: 10.1097/01.blo.0000093004.90435.d1. PMID 14646749
- [Result] Johnson TC, Tatman PJ, Mehle S, Gioe TJ. Revision surgery for patellofemoral problems: should we always resurface? Clin Orthop Relat Res. 2012 Jan;470(1):211-9. doi: 10.1007/s11999-011-2036-2. PMID 21858641
- [Result] Gioe TJ, Sharma A, Tatman P, Mehle S. Do "premium" joint implants add value?: analysis of high cost joint implants in a community registry. Clin Orthop Relat Res. 2011 Jan;469(1):48-54. doi: 10.1007/s11999-010-1436-z. PMID 20568026